CLINICAL TRIAL: NCT03523663
Title: Algorithm to Quantitatively Determine the Ideal Drug Dose to Treat Attention Deficit Hyperactivity Disorder
Brief Title: System for Determining Ideal Drug Doses for ADHD - Stages 1 and 2
Status: Terminated | Type: Observational
Why Stopped: difficulty recruiting pediatric participants followed by a prolonged shut down due to COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0857; A536200 (Other: UW Madison); SMPH\DPT NEUROSCIENCE (Other: UW Madison); Protocol Version 8/1/2019 (Other: UW Madison)
Record Dates: First submitted 2016-01-06; First posted 2018-05-14 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: healthy children without ADHD or other mental health issues
  Interventions: Other: no intervention. measure eye movement data
- ADHD: children diagnosed with ADHD
  Interventions: Other: no intervention. measure eye movement data

INTERVENTIONS:
Other: no intervention. measure eye movement data

SUMMARY:
The goal of this study is to create a formal, quantitative methodology to determine what is the most beneficial dose of Central Nervous System (CNS) stimulant (Ritalin, methylphenidate) to improve cognitive and behavioral function of children diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) individually. If successful, it will change the way in which the dose of CNS stimulant for treating ADHD is determined for children in need of therapeutic intervention. The project will be focused on developing the necessary methodology to analyze the children's data with the drift-decision model (DDM), and to develop the required technology, i.e., a computer game with which to measure cognitive/behavioral function and its validation with eye-tracking measurements.

ELIGIBILITY:
Inclusion Criteria:

* 8-12 years of age;
* Accompanied by caregiver (parent or legal guardian);
* Able to understand and speak English;
* Able to read basic English;
* No counseling or current/past history of psychiatric illness, as confirmed by the Child Behavior Checklist (CBCL) and Conner's rating scale

Exclusion Criteria:

* Active psychosis or suicidality
* History of primary psychotic disorder (e.g., schizophrenia) or bipolar disorder
* Recent (past 2 weeks) substance abuse or dependence
* History of brain damage or significant developmental delay
* Unstable medical condition such as newly diagnosed Type I Diabetes or Rheumatoid arthritis
* Use of oral steroids
* Participation in the last 30 days in a clinical study involving an investigational drug
* Current use of a psychotropic medicine

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-01; Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Task choice | At the time of testing (the investigators are measuring acute effects, not following outcomes based on a treatment)
  Subjects will perform different cognitive tasks and we will record their choices.
Reaction time | At the time of testing (the investigators are measuring acute effects, not following outcomes based on a treatment)
  The investigators record how long it took them to make their choices.
Eye position | At the time of testing (the investigators are measuring acute effects, not following outcomes based on a treatment)
  The tasks are eye movement based. The investigators record where the subjects were looking as voltages, which are converted to x/y coordinates through a calibration, throughout the different events of the task.

CONTACTS AND LOCATIONS:
Overall Officials: Luis C Populin, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Wisconsin Institutes of Medical Research, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No